CLINICAL TRIAL: NCT01477879
Title: Phase II Clinical Trial of Versabase/Sarracenia Purpurea Versus Placebo
Brief Title: Hsv 1 and 2 Gowey Protocol Versus Placebo
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Naturopaths International (Other)
Responsible Party: Principal Investigator, Dr. Brandie Gowey, NMD, Brandie Gowey, Naturopaths International
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSV1&2
Record Dates: First submitted 2011-11-15; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Herpes
MeSH Terms: conditions — Herpes Simplex | interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Versabase/20% S. purpurea extract (Active Comparator)
  Interventions: Other: Versabase gel with sarracenia purpurea 20% liquid extract
- placebo (versabase gel only) (Placebo Comparator): placebo used will be versabase gel alone
  Interventions: Other: placebo (versabase gel only)

INTERVENTIONS:
Other: Versabase gel with sarracenia purpurea 20% liquid extract — Topical application of gel/plant mix to lesions
  Arms: Versabase/20% S. purpurea extract
Other: placebo (versabase gel only) — versabase gel only
  Arms: placebo (versabase gel only)

SUMMARY:
This study will compare efficacy of versabase gel with 20% sarracenia purpurea versus placebo applied every 3-4 hours to herpes lesions.

DETAILED DESCRIPTION:
Patients screened for hsv one or two. Patients with herpes given a 1/8 oz of gel. Researcher does not know which is active and which is placebo (placebo is actually just versabase gel). Patent applies gel to lesions every 3-4 hours. Returns to clinic on days 3, 5, and 14 for evaluation. Up to 50 patients may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

- Hsv 1&2

Exclusion Criteria:

* No active lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pain | 2 weeks
  Pain scale-- subjective
Size | 2 weeks
  Measure lesion size over 2 weeks

SECONDARY OUTCOMES:
Appearance | 2 weeks
  Photo taken of lesion w patient informed consent

CONTACTS AND LOCATIONS:
Locations (1):
- Naturopaths international, Flagstaff, Arizona, United States